CLINICAL TRIAL: NCT05325190
Title: Efficacy and Safety of Granisetron Transdermal Patch System for Prevention of Chemotherapy-induced Delayed Nausea and Vomiting by CapeOX：A Single-Arm, Open-Label, Phase II Study.
Brief Title: Granisetron Transdermal Patch System for Prevention of CINV by CapeOX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: E20210665A
Record Dates: First submitted 2022-03-27; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-03

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Granisetron

STUDY DESIGN:
Intervention Model Description: Granisetron transdermal patch for the prevention and treatment of CINV
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Granisetron transdermal patch 3.1mg was given 48 hours before the first day of chemotherapy, Dexamethasone 12mg was taken orally on the first day of chemotherapy and dexamethasone 8mg was taken orally on the second and third days of chemotherapy,3.1mg granisetron transdermal patch was replaced on the 5th day of chemotherapy. Granisetron transdermal patch was removed and discarded on the 12th day of chemotherapy.
  Interventions: Drug: Granisetron Transdermal Patch System

INTERVENTIONS:
Drug: Granisetron Transdermal Patch System — Granisetron transdermal patch 3.1mg was given 48 hours before the first day of chemotherapy, Dexamethasone 12mg was taken orally on the first day of chemotherapy and dexamethasone 8mg was taken orally on the second and third days of chemotherapy,3.1mg granisetron transdermal patch was replaced on the 5th day of chemotherapy. Granisetron transdermal patch was removed and discarded on the 12th day of chemotherapy.
  Other Names: Sancuso®

SUMMARY:
This study aims to explore the prevention of delayed chemotherapy induced by CAPOX regimen with granisetron transdermal patch。

DETAILED DESCRIPTION:
Chemotherapy induced nausea and vomiting (CINV) is one of the most common side effects of tumor chemotherapy. Anorexia occurs in mild cases, electrolyte and acid-base balance disorders and malnutrition even occur in severe cases. Some patients will also have anxiety, fear and depression, which seriously affect the quality of life. This study explored the efficacy and safety of granisetron transdermal patch in the prevention of delayed nausea and vomiting caused by capeox chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged >18 years.
* Eligible patients were diagnosed with a colorectal malignancy and scheduled to receive chemotherapy of CapeOx regimens.
* The Eastern Cooperative Oncology Group Performance Status (ECOG PS) scores of patients were between 0 and 2.
* Patients with life expectancy≥6 months.
* Patients with the ability to understand the study and are willing to sign written informed consent document.
* Patients who were able to read, understand and follow the study procedures，and completed the questionnaire unaided.

Exclusion Criteria:

* Patients with metabolic and haematological abnormalities who are unsuitable for chemotherapy. The following criteria are included: (1) Abnormal of blood routine: absolute neutrophil count(ANC) <1.5*109/L，white blood cell count (WBC)<3.0*109/L, platelet count (PLT) <100*109/L or hemoglobin (HB)<100g/L;(2) Abnormal liver function: aspartate aminotransaminase (AST) and/or aspartate aminotransferase (ALT)≥2.5*ULN, bilirubin is greater than 1.5 times the upper limit of normal value (ULN). In patients with known liver metastasis: AST is greater than or equal to 5 times the upper limit of normal value (ULN); ALT is greater than or equal to 5 times the upper normal value (ULN); (3) Abnormal renal function: serum creatinine is greater than 1.5*ULN.
* Patient had symptomatic primary or metastatic central nervous system malignancies.
* Patient used any drug with potential antiemetic effect within 7 days before receiving chemotherapy: 5-HT3 receptor antagonist (such as granisetron), phenothiazide (such as chlorpromazine), phenylbutanone (such as haloperidol), benzamide (such as metoclopramide), domperidone, cannabinoids, herbal medicine with potential antiemetic effect, anisodamine, seclizine, etc.
* Patients began to receive benzodiazepines or opioids within 48 hours before the first day of the study (except for single daily use of triazolam, temazepam or midazolam).
* Patients shall not receive any dose of systemic glucocorticoid treatment within 72 hours before the first day, except as specified in the protocol.
* Patients with historical or predisposing cardiac conduction abnormalities (such as torsade de pointe, ventricular tachycardia, long QT interval syndrome, or others), excluding incomplete right bundle branch block.
* Patients with severe cardiovascular diseases include acute myocardial infarction, unstable angina pectoris, significant membranous or pericardial disease, history of ventricular tachycardia, symptomatic chronic heart failure (New York Heart Association [NYHA] class III-IV) and uncontrolled hypertension.
* Patients with severe emotional or mental disorders.
* Patients are taking or has used the following CYP3A4 inducers within 30 days before the first day of treatment, which will affect the efficacy of therapeutic drugs according to the evaluation of the researcher.
* Patients are taking or has used the following CYP3A4 substrates and inhibitors within 7 days before the first day of treatment, which will significantly increase the adverse events related to therapeutic drugs according to the evaluation of the investigator.
* Patients with active phase infection (e.g. pneumonia) or any uncontrolled disease (such as diabetic ketoacidosis or gastrointestinal obstruction), researchers believe that treatment may confuse research results or lead to uncertainty risk.
* Pregnant women, lactating women, or women of childbearing age with positive blood and/or urine HCG test results before the test. Male and female subjects did not take effective contraceptive measures, or planned to be pregnant within 6 months after the start of the trial.
* Patients have any medical history that the investigator believes may confound the results of the study or expose the patient to unnecessary risks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2021-10-10 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Complete control rate of delayed nausea and vomiting | 24 hours to 20 days before the first day of chemotherapy
  Complete control rate of delayed nausea and vomiting (CC, 24 hours to 20 days before the first day of chemotherapy)

SECONDARY OUTCOMES:
Dates of delayed complete control | from 24 hours to the 20th day of chemotherapy
  Definition of DDCC (dates of delayed complete control): from 24 hours to the 20th day of chemotherapy, the patient has no vomiting, no rescue treatment, no nausea (VAS < 5mm) or mild nausea (VAS < 25mm, mild);
Complete control rate of acute nausea and vomiting | 24 hours to 20 days before the first day of chemotherapy
  From 0 hour to 24 hours after chemotherapy, the patients did not vomit or need rescue treatment, and there was no incidence of nausea (VAS < 5mm) or mild nausea (VAS < 25mm).
Proportion of subjects receiving remedial treatment | 24 hours to 20 days before the first day of chemotherapy
  The investigator evaluated the degree of nausea and vomiting reported by the patient and the observed clinical manifestations according to the study
  In the judgment of the patient, remedial treatment can be used only when necessary to treat nausea or vomiting, and remedial treatment shall not be used when the patient does not have such symptoms.
Changes of FLIE score before and after treatment | 24 hours to 20 days before the first day of chemotherapy
  FLIE includes 9 questions about nausea and 9 questions about vomiting. The answers to each item were marked according to the visual analog scale with a score of 7. The nausea score, vomiting score and total score were calculated by summing the answers of each category and the total answer. Considering the purpose of this scheme, "no impact" on daily life is defined as that the average item score is greater than 6 points (total score > 108) according to 7 subscales.
Changes of hospital anxiety and Depression Scale (HAD) scores before and after treatment | 24 hours to 20 days before the first day of chemotherapy
  HAD is mainly used for screening anxiety and depression of patients in general hospitals. There are 14 items in this scale, including 7
  Depression was assessed in items (21 points in total), and anxiety was assessed in 7 items (21 points in total). The score of depression subscale is 0-7, indicating no symptoms; 8-10 points are suspicious of depressive symptoms, and 11-21 points must have depressive state. Anxiety subscale score 0-7
  Asymptomatic; The anxiety symptoms are suspicious on 8-10 points, and there must be anxiety on 11-21 points.

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by NCI CTC AE V5.0. | 24 hours to 20 days before the first day of chemotherapy
  Number of participants with treatment-related adverse events as assessed by NCI CTC AE V5.0 were recorded at any time, and the patients were followed up until death.

CONTACTS AND LOCATIONS:
Overall Officials: Cong Wang, Doctor, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang C, Jiang Z, Zhang J, Zhuang Y, Sun L, Zhang J, Quan M, Lan L, Li Y, Wang B, Pan Z, Yan Z. Prolonged administration of the granisetron transdermal delivery system reduces capecitabine plus oxaliplatin regimen induced nausea and vomiting. BMC Cancer. 2024 Jul 18;24(1):867. doi: 10.1186/s12885-024-12616-9. PMID 39026165